CLINICAL TRIAL: NCT05376657
Title: Evaluation of Antioxidant and Skin Beauty Effects of Cherry Collagen Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 22-010-B
Record Dates: First submitted 2022-05-12; First posted 2022-05-17 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Skin Condition
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo drink
- Cherry collagen drink (Experimental)
  Interventions: Dietary Supplement: Cherry collagen drink

INTERVENTIONS:
Dietary Supplement: Cherry collagen drink — consume 1 sachet per day
  Other Names: YOUNIQUE DAILY YOU liquid collagen shot
  Arms: Cherry collagen drink
Dietary Supplement: Placebo drink — consume 1 sachet per day
  Arms: Placebo drink

SUMMARY:
To assess cherry collagen drink on skin condition improvement

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, liver, kidney.
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* Received facial laser therapy, chemical peeling or UV overexposure (> 3 hr/week) in the past 4 weeks.
* Constant drug use
* Students who are currently taking courses taught by the principal investigator of this trial.
* Body weight < 50 kg.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-09-03 (Actual)

PRIMARY OUTCOMES:
The change of skin wrinkles | Change from Baseline skin wrinkles at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin wrinkles. Units: arbitrary units
The change of skin texture | Change from Baseline skin texture at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin texture. Units: arbitrary units
The change of skin collagen density | Change from Baseline skin collagen density at 8 weeks
  DermaLab® Series SkinLab Combo was utilized to measure skin pores. Units: arbitrary units
The change of skin elasticity | Change from Baseline skin elasticity at 8 weeks
  Soft Plus was utilized to measure skin elasticity. Units: arbitrary units

SECONDARY OUTCOMES:
The change of skin melanin index | Change from Baseline skin melanin index at 8 weeks
  Soft Plus was utilized to measure skin melanin index. Units: arbitrary units
The change of skin L* value | Change from Baseline L* value at 8 weeks
  Chroma Meter MM500 was utilized to measure skin L* value. Units: arbitrary units, 0-100
The change of skin moisture | Change from Baseline skin moisture at 8 weeks
  Corneometer® CM825 was utilized to measure skin moisture. Units: arbitrary Corneometer® units 0-120
The change of skin spots | Change from Baseline skin spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin spots. Units: arbitrary units
The change of skin UV spots | Change from Baseline skin UV spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin UV spots. Units: arbitrary units
The change of skin brown spots | Change from Baseline skin brown spots at 8 weeks
  VISIA Complexion Analysis System was utilized to measure skin brown spots. Units: arbitrary units
The change of SOD-RBC of blood | Change from Baseline SOD-RBC at 8 weeks
  Venous blood was sampled to measure SOD-RBC
The change of t-GSH of blood | Change from Baseline t-GSH at 8 weeks
  Venous blood was sampled to measure t-GSH
The change of GST-RBC of blood | Change from Baseline GST-RBC at 8 weeks
  Venous blood was sampled to measure GST-RBC
The change of blood total antioxidant capacity (TAC) | Change from Baseline TAC at 8 weeks
  Venous blood was sampled to measure concentrations of TAC
The change of desmosine of blood | Change from Baseline desmosine at 8 weeks
  Venous blood was sampled to measure concentrations of desmosine
The change of TNF-alpha of blood | Change from Baseline TNF-alpha at 8 weeks
  Venous blood was sampled to measure concentrations of TNF-alpha
The change of transepidermal water loss (TEWL) | Change from Baseline TEWL at 8 weeks
  Tewameter® TM300 was utilized to measure TEWL. Units: g/hm²

OTHER OUTCOMES:
The change of liver function biomarkers (AST, ALT) of blood | Change from Baseline liver function biomarkers at 8 weeks
  Venous blood was sampled to measure liver function biomarkers
The change of renal function biomarkers (creatinine, BUN) of blood | Change from Baseline renal function biomarkers at 8 weeks
  Venous blood was sampled to measure renal function biomarkers
The change of self-assessment skin condition | Change from Baseline skin condition at 8 weeks
  A self-assessment questionnaire was collected to evaluate skin condition

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hua Liang, Principal Investigator — Chia Nan University of Pharmacy ＆ Science
Locations (1):
- Chia Nan University of Pharmacy & Science, Tainan, Taiwan